CLINICAL TRIAL: NCT05903911
Title: Trans Care: An Online Intervention to Reduce Symptoms of Gender Dysphoria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-0644: RCT; UW Baldwin Endowment (Other: UW Madison); A171600 (Other: UW Madison); Protocol Version 10/17/24 (Other: UW Madison)
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Intervention Model Description: 130 participants randomized to intervention and 130 to waitlist control
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans Care Intervention (Experimental)
  Interventions: Other: Trans Care Web App
- Waitlist Control (No Intervention)

INTERVENTIONS:
Other: Trans Care Web App — an educational and interactive website designed to improve coping strategies of TNB individuals
  Arms: Trans Care Intervention

SUMMARY:
The current project aims to improve the well-being of trans and nonbinary (TNB) individuals through an online intervention (Trans Care) targeting the reduction of symptoms of gender dysphoria. The Trans Care intervention will involve the creation of an online intervention comprised of eight modules intended to reduce symptoms of gender dysphoria, increase active coping, and improve the well-being of TNB individuals. Aim 2 is a randomized controlled trial of the proposed intervention and will enroll 260 TNB participants.

DETAILED DESCRIPTION:
The overall purpose of this project is to create a free intervention that can be disseminated widely throughout TNB communities to improve well-being in an easy, accessible way. Development and execution of the Trans Care intervention involves two primary aims:

* Aim 1) Feasibility and acceptability analysis (FAA) [represented by NCT05884307]
* Aim 2) A pilot randomized controlled trial (RCT) of Trans Care's efficacy [represented in this study record]

Aim 2 is a RCT in which participants' scores of psychological wellbeing and coping strategies in the intervention vs waitlist control group will be analyzed. Additionally, participants who drop out of the RCT will be asked to complete measures at dropout to determine what dose size of Trans Care (i.e., how many modules) is necessary to have a significant change in mental well-being. Finally, waitlisted participants will be offered the intervention within one month of the completion of data collection.

Aim 2 Hypotheses:

* TNB Participants who received the Trans Care intervention will demonstrate improvement on quantitative measures of psychological well-being, GD symptoms, and coping strategies compared to waitlisted individuals.
* Changes will be maintained at 3 months follow-up indicating that the Trans Care intervention has a sustained impact on improving TNB individuals' coping.

Aim 2 Endpoints:

The primary endpoint of Aim 2 will be to determine if participants who engaged the Trans Care intervention experienced psychological improvement in their mental health as a result of completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Identify as transgender, transsexual, nonbinary, and/or have a transgender history.
* Experience gender dysphoria.
* Time available to commit to completing a 4-5-hour online intervention and 1-2 hours to complete follow up surveys

Exclusion Criteria:

* under 18 years old
* individual does not identify as transgender, transsexual, nonbinary, and/or have a transgender history
* does not experience gender dysphoria
* is unable to commit to the time requirements of the study
* does not have access to an internet compatible device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety, and Stress Scale (DASS-21) Score | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  DASS-21 is a composite measurement used to assess symptoms of depression, anxiety, and stress in community settings. The 21-item survey is comprised of three subscales for Depression, Anxiety, and Stress. Responses are provided on a 4-point Likert scale, Where 0 = Did not apply to me, 1 = applied to me some degree, or some of the time, 2 = applied to me a considerable degree or good part of time, and 3 = applied to me very much or most of the time. Total possible range of scores is from 0 to 63, with higher scores indicating higher levels of symptoms.
Change in Gender Congruence and Life Satisfaction Scale (GCLS) Score | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  GCLS measures gender congruence and life satisfaction in a 38-item self assessment, for a total possible range of scores from 38-190 where higher values indicate greater gender congruence, greater gender-related well-being, and greater life satisfaction.
Change in Modified Gender Minority Stress and Resilience measure (M-GMSRM) Score | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  Total scores are calculated for each scale based on summed values assigned to possible response options. The first 8 items are scored 0 for "never," 1 for "yes, before age 18," 2 for "yes, after age 18," and 3 for "yes, in the past year." Scores from these items are then summed where a higher score indicates more frequent and recent experiences of gender related prejudice. All other items are scored from 0 - 4 according to responses ranging from strongly disagree to strongly agree. Items within each subscale (i.e., non-affirmation of identity, internalized transphobia, and negative expectations for the future) are summed with high scores indicating greater distress.
Change in Trans and Nonbinary Coping Measure (TNCM) Score | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  TNCM assesses the unique ways of coping with gender-related stress. The measure includes six subscales (Social Support/Connection (5 items); Social Activism (4 items); Hope (5 items); Strategic Gender Expression (5 items); Behavioral Avoidance (5 items); Identity Nondisclosure (4 items). Responses to items are recorded on a 5-point scale from 1 (I do not do this) to 5 (I almost always do this). Scale items are summed to create subscale scores. A higher score indicates greater frequency of use of that coping strategy.
Alcohol Use Disorder Identification Test | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  This is scored from 0-4 where higher scores are indicative of increased dependence on alcohol.
Number of Days in the Past Week You Consumed Alcohol | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  7 = 7 days, 6 = 6 days, 5 = 5 days, 4 = 4 days, 3 = 3 days, 2 = 2 days, 1 = 1 day, 0 =no days
Quantity of Alcohol Use | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  How many alcoholic drinks, on average, have you had per day during the pastweek? An alcoholic drink is defined as 1 beer, 1 glass of wine, 1 shot of alcohol, or 1mixed drink.
  Response options:
  5 = 12+ drinks, 4 = 8-11 drinks, 3 = 5-7 drinks, 2 = 3-4 drinks, 1 = 1-2 drinks, 0 =none
Change in Multidimensional Gender Dysphoria Measure Scores | before and after intervention (participants will have up to 1 month to complete intervention), 3 month follow up
  The Multidimensional Gender Dysphoria Measure is a 25-item survey each scored from 1 (strongly disagree) to 6 (strongly agree) for a total possible range of scores of 5-30 in each of 5 domains: Body Gender Dysphoria, Social Gender Dysphoria, Variability of Gender Dysphoria, Relief from Gender Dysphoria, and Internalized Gender Normativity. Higher scores indicate greater gender dysphoria distress.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Budge, PhD, LP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindley, L., & Budge, S. L. (2022). Development and validation of the Trans and Nonbinary Coping Measure (TNCM): A measure of trans and nonbinary specific ways of coping with gender-related stress. Psychology of Sexual Orientation and Gender Diversity. Advance online publication. https://doi.org/10.1037/sgd0000618
- See also: Public Record for Trans Care: An Online Intervention to Reduce Symptoms of Gender Dysphoria Feasibility and Acceptability Study — https://clinicaltrials.gov/ct2/show/NCT05884307